CLINICAL TRIAL: NCT06332885
Title: Zephyr Valve Japan Post-Marketing Surveillance
Status: Recruiting | Type: Observational
Sponsor: Pulmonx Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 630-2001-01
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Emphysema; COPD; Severe Emphysema
Keywords: Bronchoscopic lung volume reduction; Zephyr Valves
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Single Group Assignment: Bronchoscopic lung volume reduction with Zephyr Valves
  Interventions: Device: Zephyr Endobronchial Valve

INTERVENTIONS:
Device: Zephyr Endobronchial Valve — Zephyr Valve provides an alternative technique to achieve bronchoscopic lung volume reduction (BLVR) using a minimally invasive approach. Zephyr Valve is a tiny unidirectional valve. During BLVR, multiple valves are placed to occlude a hyperinflated lobe of the lungs, allowing air to escape while blocking airflow into the treated lobe. This is intended to result in a reduction in lung volume and hyperinflation in the targeted area. Consequently, the remaining lobes can expand more fully, the overall lung works more efficiently, with resultant improvement in overall lung function in patients with hyperinflation associated with severe emphysema.

SUMMARY:
This is a multicenter, prospective, observational surveillance enrolling 140 consecutive patients with severe emphysema who are candidates for bronchoscopic lung volume reduction using Zephyr Endobronchial Valve at up to 20 centers across Japan and followed for 12 months.

DETAILED DESCRIPTION:
This is a multicenter, prospective, observational surveillance across 20 centers in Japan enrolling 140 consecutive adult patients with hyperinflation of the lungs due to severe emphysema who are considered to be appropriate candidates for BLVR using Zephyr Endobronchial Valve (EBV, Pulmonx Corporation) and confirmed to have little to no collateral ventilation in the target lobe.

Enrolled (consented) subjects will undergo a bronchoscopy procedure with the Chartis assessment to confirm that little to no collateral ventilation is present (CV- status) followed by EBV placement in the most diseased lobe. Subject will be hospitalized for a minimum of 3 nights for observation and followed up for 12 months.

Subjects with collateral ventilation will be exited from the surveillance without treatment.

The primary endpoint is incidence rate of pneumothorax at Day 45 post-index procedure.

The effectiveness will be evaluated from Baseline to specified timepoint based on changes in lung function, exercise capacity, dyspnea and quality of life. A high-resolution computed tomography (HRCT) will be performed at Day 45 and Month 12 to determine Treated Lobe Volume Reduction (TLVR). Lung function will be assessed at Month 3, 6 and 12 by measuring post-bronchodilator forced expiratory volume in 1 second (FEV1), residual volume (RV) and 6 Minutes Walking Distance. The safety will be evaluated based on incident rate of treatment emergent adverse events through Month 12.

Subjects will be required to complete a pulmonary rehabilitation program between Day 45 and Month 3 per local/national guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is deemed eligible for BLVR using Zephyr Valve, as determined by their treating physician in accordance with Japanese guidelines and approved instruction for use. These include:

   * Recent respiratory rehabilitation completed within the last 6 months
   * Not actively smoking (for at least 4 months)
   * TLC ≥ 100%
   * RV ≥ 175%
   * FEV1 15-45% post-bronchodilator
   * 6MWD 100-500 m
   * mMRC score ≥ 2
   * No coagulation disorder
   * No evidence of active respiratory infection
2. Patient has little to no collateral ventilation (CV-) between the target and ipsilateral lobe as confirmed by Chartis prior to undergoing BLVR.
3. Patient is willing and able to provide informed consent to allow data collection.

Exclusion Criteria: None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The surveillance population will be adult patients (18 years or older) in Japan with hyperinflation of the lungs due to severe emphysema who are considered by their treating physician to be appropriate candidates for BLVR using Zephyr Valve and confirmed to have little to no collateral ventilation (CV-) in the target lobe. The surveillance will enroll all patients treated at the participating hospitals who provide written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of pneumothorax at 45-days post-Zephyr Valve index procedure. | 45-days post-Zephyr Valve index procedure
  The percentage of study subjects who experience pneumothorax within 45-days post-Zephyr Valve index procedure.

OTHER OUTCOMES:
Forced Expiratory Volume in 1 second (FEV1) | Month 3, 6, 12
  The volume of air in liters exhaled in the first second during forced exhalation after maximal inspiration. The MCID is a volume increase by at least 12%.
Residual Volume (RV) | Month 3, 12
  The volume of air in remaining in the lungs after maximum forceful expiration. The MCID is a decrease by at least 310 mL.
Treated lobe volume reduction (TLVR) | Day 45, Month 12
  Treated lobe volume reduction is determined by HRCT and measured from Baseline to a given timepoint in mL and percentage of subjects achieving a ≥ 350 mL decrease
Six-Minute Walk Distance (6MWD) | Month 3, 6, 12
  Measures the distance (in m) an individual is able to walk over a total of 6 minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in 6 minutes. The MCID is an increase of 6MWD by at least 26 m.
Modified Medical Research Council Dyspnea (mMRC) Scale score | Month 3, 6, 12
  A self-rating tool to measure the degree of disability that breathlessness poses on day-to-day activities on a scale from 0 to 4 as follows:
  * 0: Dyspnea only with strenuous exercise
  * 1: Dyspnea when hurrying or walking up a slight hill
  * 2: Walks slower than people of same age because of dyspnea or has to stop for breath when walking at own pace
  * 3: Stops for breath after walking 100 yards (91 m) or after a few minutes
  * 4: Too dyspneic to leave house or breathless when dressing The MCID is a total score reduction by at least 1 point.
St. George's Respiratory Questionnaire (SGRQ) Total Score | Month 3, 6, 12
  A validated, disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease. Total score for 3 component domains (impact, activity, symptoms) ranges from 0 to 100. Higher score indicates worse quality of life. The MCID is a decrease by at least 4 points.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Melloy, MBA, Study Director — Pulmonx Corporation
Locations (17):
- Japan (17):
  - Tosei General Hospital, Aichi
  - Gifu Prefectural Medical Center, Gifu
  - Kanagawa Cardio Chest Center, Kanagawa
  - Kanazawa University Hospital, Kanazawa
  - St Marianna University Hospital, Kawasaki
  - Matsusaka Civic Hospital, Mie
  - Nagasaki University Hospital, Nagasaki
  - Nagoya Medical Center, Nagoya
  - Okayama Medical Center, Okayama
  - Kinki Chuo Chest Medical Center, Osaka
  - Hokkaido University Hospital, Sapporo
  - Tohoku University Hospital, Sendai
  - Shiga University Hospital, Shiga
  - Tokyo National Hospital, Tokyo
  - Fujita Health University Hospital, Toyoake
  - Dokkyo University Hospital (Pulmonary Medicine and Clinical Immunology), Utsunomiya
  - Dokkyo University Hospital, Utsunomiya

IPD SHARING:
Plan to Share IPD: No
All data will be aggregated and analyzed. No IPD will be made available for sharing to other researchers.